CLINICAL TRIAL: NCT05608876
Title: A Phase II, Open Label, Single Arm Study To Assess The Efficacy Of Intratumoral Tigilanol Tiglate In Various Head And Neck Solid Malignancies
Brief Title: A Clinical Study to Investigate the Efficacy of Tigilanol Tiglate Directly in Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QBiotics Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QB46C-H08; U1111-1282-3152 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2022-10-16; First posted 2022-11-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Squamous cell carcinomas; Sino-nasal cancers; Salivary gland cancers; Peri-stomal laryngeal carcinomas
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Salivary Gland Neoplasms | interventions — EBC-46

STUDY DESIGN:
Intervention Model Description: Open label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm, Open Label (Experimental): Single or multiple Intratumoural injections of tigilanol tiglate at up to a fixed dose of 3.6 mg/m2 (Body Surface Area [BSA]) per treatment.
  Interventions: Drug: Tigilanol Tiglate

INTERVENTIONS:
Drug: Tigilanol Tiglate — Tigilanol tiglate is a novel, short-chain diterpene ester in clinical development for intratumoural treatment of a wide range of solid tumours.
  Other Names: EBC-46

SUMMARY:
A Phase II, open label, single arm study to assess the efficacy of intratumoural tigilanol tiglate in various head and neck solid malignancies.

DETAILED DESCRIPTION:
Primary Objective

1. To evaluate tumour ablation following treatment(s) with intratumoural injections of tigilanol tiglate.

Secondary Objectives

1. To assess the safety and tolerability of intratumoural injections with tigilanol tiglate.
2. To evaluate disease control by assessing time to local disease recurrence from last treatment.
3. To evaluate the tumour recurrence rate at injected tumour sites.
4. To evaluate survival by assessing Progression Free Survival (PFS).

Exploratory Objectives

1. To assess the impact on Quality of Life (QoL).
2. To assess the degree of wound healing after each treatment.
3. To assess the tumour response in injected and non-injected tumours, based on Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
4. To assess the tumour response according to intratumoural Response Evaluation Criteria in Solid Tumours (itRECIST).
5. To assess changes in tumour biomarkers.
6. To assess the tumour microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Are willing and able to provide written informed consent for the study prior to any protocol-specific procedures and to comply with all local and study requirements.
2. Are ≥ 18 years of age on the day of providing informed consent.
3. Have a histologically confirmed diagnosis of a solid head and neck malignancy and have either recurrent disease and/or metastatic disease, or have failed on at least one line of systemic therapy. Tumour types can include: HNSCC, sino-nasal cancers, salivary gland cancers, and peri-stomal laryngeal carcinomas with pre-existing tracheostomy.
4. Have disease that is amenable to intratumoural injection either by palpation or under ultrasound guided injection. Lymph nodes with metastatic disease from the patient's head and neck cancer can be selected for treatment. Note: Measurable disease as per RECIST v1.1. is not mandatory.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
6. Have life expectancy of more than 12 weeks.
7. Female participants who are Women of Child-Bearing Potential (WOCBP) must have a negative serum pregnancy test at Screening (within 14 days of the first study drug administration), must be willing to use a highly effective contraception from date of consent, throughout the study period and up to 30 days after the last study drug administration, and must not be breastfeeding.
8. Male participants with a potentially fertile female partner are eligible if they have had a vasectomy or are willing to use adequate contraception from prior to commencement of study drug administration, throughout the study period and up to 30 days after the last study drug administration, and must not donate sperm throughout the study period and up to 30 days after the last study drug administration.

Exclusion Criteria:

1. Are planning to receive intratumoural treatment or radiotherapy to any of the tumours intended for injection within 28 days prior to Screening, or during treatment with tigilanol tiglate.
2. Have a tumour intended for injection that is immediately adjacent to, or with infiltration into, any major artery or vein (e.g., if the tumour for injection is located adjacent to the jugular vein).
3. Have a tumour intended for injection located in an area where post-injection swelling could compromise the airway.
4. Have a tumour intended for injection that is a nasal tumour extending into the Ethmoid sinus.
5. Have had any previous intervention (extensive surgery or radiation therapy) in the area of a tumour intended for injection that is in proximity of the airway (such that tracking of the injected fluid may be unpredictable and could lead to airway swelling). Patients with a permanent tracheostomy can be included.
6. Are receiving or have received other investigational agents or have used an investigational device without undergoing a 28-day (or 5 half-lives, whichever is shorter) wash-out period prior to their first treatment with tigilanol tiglate. These patients must have recovered from all AEs due to previous investigational therapies to ≤ Grade 1 at baseline.
7. Are receiving or have received systemic anticancer therapy, or therapeutic radiation treatment, without undergoing a 28-day (or 5 half-lives, whichever is shorter) wash-out period prior to their first treatment with tigilanol tiglate. These patients must have recovered from all AEs due to previous therapies to ≤ Grade 1 at baseline.
8. Have had major surgery within 28 days of their first treatment with tigilanol tiglate or anticipate the need for major surgery during the study period. Minor surgical procedures are permitted, but with sufficient time for wound healing.
9. Have known, current or history of active cerebral metastasis and/or carcinomatous meningitis.
10. Have any bleeding diathesis or coagulopathy that would make intratumoural injection or biopsy unsafe, or if they are on therapeutic warfarin therapy.
11. Have a history of allergic reactions or severe hypersensitivity (Grade ≥ 3) attributed to tigilanol tiglate or compounds of similar chemical or biologic composition to tigilanol tiglate, any of its excipients or other agents used in the study.
12. In the opinion of the treating Investigator, the patient is not an appropriate candidate for the study for any reason (e.g., they have a known psychiatric or substance abuse disorder that would interfere with their ability to cooperate with the requirements of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Tumour Response | 72 weeks
  Proportion of participants who have achieved partial or complete ablation of treated tumour(s) and/or tumour segment(s) following injection(s) with tigilanol tiglate.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 72 weeks
  Total number of Adverse Events (AEs) and Serious Adverse Events (SAEs) and number of AEs and SAEs deemed related to tigilanol tiglate.
Disease Control | 72 weeks
  Time from last treatment to recurrence of disease at injection site(s).
Local Recurrence Rate at injection site(s) | 6-, 12-, and 18-months after first treatment.
  Percentage of participants with local recurrence at injection site(s) at 6-,12- and 18-months after first treatment.
Progression Free Survival (PFS) | 72 weeks
  Progression Free Survival (PFS) based on RECIST v1.1 defined as the length of time between first treatment and the date of the first occurrence of disease progression.

OTHER OUTCOMES:
General Cancer Quality of Life (QoL) Assessment | 72 weeks
  Quality of Life will be assessed via The European Organisation for Research and Treatment of Cancer (EORTC) general cancer specific questionnaire (QLQ-C30).
  For the QLQ-C30 all of the scales and single-item measures range in score from 0 to 100. A high scale score will represent a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/QoL represents a high quality of life, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Head and Neck Cancer Quality of Life (QoL) Assessment | 72 weeks
  Quality of Life will also be assessed via The European Organisation for Research and Treatment of Cancer (EORTC) questionnaire designed to assess the quality of life of head and neck cancer patients (QLQ-H&N35).
  For the QLQ-H&N35, all of the scales and single-item measures range in score from 0 to 100. For all the scales and single-items a high score represents a high level of symptomatology or problems.
Wound Healing | 72 weeks
  Degree of wound healing at injection site(s) will be assessed using a specifically designed Injection Site Assessment Worksheet, observed at monthly intervals up to 72 weeks
Tumour Response Rate Of Both Injected And Non-Injected Tumours | 72 weeks
  Overall Response Rate of both injected and non-injected tumours based on RECIST v1.1.
Tumour Response Rate | 72 weeks
  Overall Response Rate based on itRECIST.
Evaluation of Peripheral Blood Mononucleocytes (PBMCs) | 24 weeks
  Evaluation of Peripheral Blood Mononucleocytes (PBMCs).
Evaluation of circulating tumour DNA (ctDNA) | 24 weeks
  Evaluation of circulating tumour DNA (ctDNA).
Tumour Microenvironment | 14 days after the first treatment.
  To assess changes in the tumour microenvironment by looking at the change from baseline of immune cell infiltration in tumour biopsy tissue collected after injection with tigilanol tiglate.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallagher, MBBS, Principal Investigator — The Kinghorn Cancer Centre; David Owens, MBchB, Principal Investigator — Cardiff and Vale University Health Board - University Hospital of Wales (UHW); Anthony Kong, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Joseph Sacco, MBchB, Principal Investigator — The Clatterbridge Cancer Centre NHS Foundation Trust; Benedict Panizza, MBBS MBA, Principal Investigator — Metro South Hospital and Health Service, via the Princess Alexandra Hospital; Kevin Harrington, BSc MBBS, Principal Investigator — Royal Marsden NHS Foundation Trust; George Mochloulis, MD CCST, Principal Investigator — East and North Hertfordshire NHS Trust (Incorporating Mount Vernon Cancer Centre) of Lister Hospital
Locations (7):
- Australia (2):
  - The Kinghorn Cancer Centre, Sydney, New South Wales
  - Metro South Hospital and Health Service, via the Princess Alexandra Hospital, Brisbane, Queensland
- United Kingdom (5):
  - Cardiff and Vale University Health Board - University Hospital of Wales (UHW), Cardiff, Cardiff
  - East and North Hertfordshire NHS Trust (Incorporating Mount Vernon Cancer Centre) of Lister Hospital, Stevenage, Hertfordshire
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - The Royal Marsden NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No